CLINICAL TRIAL: NCT01728350
Title: Improving Well-Being After TBI Through Structured Volunteer Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H133A120032-1
Record Dates: First submitted 2012-11-09; First posted 2012-11-19 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; volunteering; well being; cortisol
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Participants in this arm will participate in a novel structured volunteering intervention called HOPE - Helping Others through Purpose and Engagement. This intervention involves orientation, training, volunteer placement assistance, and problem solving and support.
  Interventions: Behavioral: HOPE - Helping Others through Purpose and Engagement
- Control (No Intervention): Participants who are randomized to the control arm will be offered the HOPE intervention at the conclusion of study.

INTERVENTIONS:
Behavioral: HOPE - Helping Others through Purpose and Engagement
  Other Names: HOPE - Helping Other through Purpose and Engagement
  Arms: Treatment

SUMMARY:
The purpose of this project is to determine if participating in volunteer activity improves the psychological well-being of individuals with traumatic brain injury (TBI).

ELIGIBILITY:
Inclusion Criteria:

* Has sustained a documented TBI that required inpatient rehabilitation;
* is at least one year post TBI;
* is age 18 or older;
* is able to commit to completing the entire three month volunteer placement;
* is English or Spanish speaking;
* receives written medical release from a physician to participate in this intervention;
* is rated a level 1-2 on the Supervision Rating Scale (functionally independent during the day);
* provides informed consent to participate

Exclusion Criteria:

* Is employed or engaged in regularly scheduled volunteer work outside of the intervention;
* obtains a score of 25 or above on the SWLS, which is 0.5 SD above the TBIMS NDB mean;
* unable to travel to assessments and placement; even with study transportation assistance;
* has been convicted of a felony, which would prohibit volunteer placement;
* unable to communicate effectively to complete standardized assessments;
* has cognitive impairment that precludes completion of baseline testing;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Satisfaction with Life Scale(SWLS)at post-intervention and follow up points. | Baseline, post-intervention, 3 mos f/u, 6 mos f/u
  A five-item, self-rated scale of global life satisfaction. Items are rated on 1-7 point Likert scale.

SECONDARY OUTCOMES:
Change from baseline on Flourishing Scale at post-intervention, and at follow-up points. | Baseline, post-intervetion, 3mos f/u, 6mos f/u
  An 8-item self-rated scale of perceived success in areas such as social relationships, self-esteem, and purpose in life. Items are rated on 1-7 point Likert scale.
Change from baseline on Brief Symptom Inventory-18(BSI-18)at post-intervention and at follow-up points. | Baseline, post-intervention, 3mos f/u, 6mos f/u
  An 18-item, self-rated measure of psychological distress. Items are rated on 0-4 Likert scale.
Change from baseline on Scale of Positive and Negative Experience (SPANE)at post intervention and at follow-up points. | Baseline, post-intervention, 3mos f/u, 6mos f/u
  A 12-item, self-rated scale that evaluates positive and negative emotions. It produces a score of positive and negative feelings that can be combined to create a balance score.
Change from baseline on Purpose in Life subscale of RyffScale of Psychological Well-Being at post-intervention and at follow-up points. | Baseline, post-intervention, 3mos f/u, 6mos f/u
  Consists of nine, self-rated items regarding individual goals, sense of direction, and meaning. This subscale was selected because volunteering has been shown to have a positive relationship with a sense of purpose in life.

OTHER OUTCOMES:
Change from baseline on Hair Cortisol test at post-intervention and at follow-up points. | Baseline, post-intervention, 3mos f/u, 6 mos f/u
  This is considered an Exploratory Measure. Cortisol has been explored as a potential biomarker of well-being; lower levels of salivary cortisol have been associated with higher levels of psychological well-being. Recently, reliable and valid methods for measuring long-term cortisol secretion through hair samples have been developed and are being used as biomarkers of chronic stress in multiple medical conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Lenore Hawley, LCSW, Principal Investigator — Craig Hospital; Lisa Payne, PhD, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States